CLINICAL TRIAL: NCT01065402
Title: A Randomized, Two-Regimen, Crossover, Comparative Study to Evaluate the Efficacy and Safety of PPB-R-203-Based Meal Versus TK9-Based Meal in 20 Patients With Diabetes
Brief Title: A Study to Evaluate the Efficacy and Safety of PPB-R-203-Based Meal Versus TK9-Based Meal in 20 Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharma Power Biotec Co., Ltd. (Industry)
Responsible Party: isRed Pharma & Biotech Research Corporation, Isredbioresearch
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: PPB-R-203-01
Record Dates: First submitted 2010-02-05; First posted 2010-02-09 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus; continuous glucose monitoring system (CGMS)
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- TK9-Based Meal (Placebo Comparator): TK9, Taikeng 9, is one commercially available rice manufacture by Yeedon Enterprise Co., Ltd. TK9-Based Meal is a diet equivalent to daily energy needs as judged by indirect calorimetry and of the same macronutrient composition.
  Interventions: Dietary Supplement: TK9-Based Meal
- PPB-R-203-Based Meal (Experimental): PPB-R-203 is manufacture by Pharma Power Biotec Co., Ltd. The composition of PPB-R-203 is resistant starch (RS). By definition, resistant starch (RS) is any starch that is not digested in the small intestine but passes to the large intestine (or the colon). Therefore, resistant starch can be regarded as a component of dietary fiber. RS intake is associated with several changes in metabolism which may confer some health benefits.
  PPB-R-203-Based is the diet equivalent to daily energy needs as judged by indirect calorimetry and of the same macronutrient composition.
  Interventions: Dietary Supplement: PPB-R-203-Based Meal

INTERVENTIONS:
Dietary Supplement: PPB-R-203-Based Meal — PPB-R-203 is manufacture by Pharma Power Biotec Co., Ltd. The composition of PPB-R-203 is resistant starch (RS). Resistant starch can be regarded as a component of dietary fiber. Some forms of RS are present naturally in many foods, and average global consumption is estimated at 3-10 g/day. PPB-R-203-Based is the diet equivalent to daily energy needs as judged by indirect calorimetry and of the same macronutrient composition.
  Arms: PPB-R-203-Based Meal
Dietary Supplement: TK9-Based Meal — TK9, Taikeng 9, is one commercially available rice manufacture by Yeedon Enterprise Co., Ltd. TK9-Based Meal is a diet equivalent to daily energy needs as judged by indirect calorimetry and of the same macronutrient composition.
  Arms: TK9-Based Meal

SUMMARY:
To evaluate the efficacy of PPB-R-203-Based Meal and TK9-Based Meal on blood glucose control in 20 patients with diabetes for 2 days.

DETAILED DESCRIPTION:
The MiniMed Medtronic CGMS (continuous glucose monitoring system), the first model approved by FDA, was used for subcutaneous glucose monitoring. The CGMS continually measures the glucose concentration of the interstitial fluid every 10 seconds and then stores an average glucose value for each 5 minutes period, for a total of up to 288 measurements each day.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus patient.
2. Aged between 20 to 65 years old.
3. Informed consent form signed.

Exclusion Criteria:

1. A recent history of drug or alcohol abuse.
2. Sensitivity to analogous product.
3. Serious cardiovascular disorders.
4. Participation in another clinical investigation study.
5. Ongoing influenza, autoimmune disease and other metabolic diseases.
6. Pregnant or lactating women.
7. Individuals are judged by the investigators or co-investigator to be undesirable as subjects.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-03 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
The daily blood glucose level will be monitored by the continuous glucose monitoring system (CGMS) device Medtronic MiniMed. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Chuang Lee Ming, Physician, Principal Investigator — National Taiwan University Hospital
Locations (1):
- PingTung Christian Hospital, Pingtung City, Taiwan